CLINICAL TRIAL: NCT06099288
Title: Strong Families Start at Home/Familias Fuertes Comienzan en Casa: A Novel Video and Motivational Interviewing Intervention to Improve Diet Quality of Low-income, Ethnically Diverse Children
Brief Title: Strong Families Start at Home/Familias Fuertes Comienzan en Casa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2022003389; R01HD108832 (NIH)
Record Dates: First submitted 2023-10-03; First posted 2023-10-25 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Metabolic Syndrome, Protection Against; Diet, Healthy
Keywords: Motivational Interview; Home-Based; Intervention; Latinx; Families; Nutrition; Cultural Tailoring; Social Cognitive Theory; Self-Determination Theory; Self-Perception Theory
MeSH Terms: conditions — Metabolic Syndrome | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: After baseline measures are complete, parent-child dyads will be randomly assigned to either the Intervention (I) or Comparison group (C) using random generator software. Because parents will need to complete a second recall over the phone after completing in-person measurements, randomization will happen over the phone. The project manager will let parents know by phone what group they are in and conduct an orientation about upcoming activities for each group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Intervention staff (Project coordinator & Community Health Workers) will know what group each participant has been allocated to. Evaluation teams will be masked. Additionally, participants will know if they have been assigned to the group focused on "child feeding" or the group focused on "child reading readiness", but will not be told that one is the intervention group and one is the comparison group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-Based Video and Motivational Interviewing Intervention (Experimental): The intervention will be delivered in English or Spanish by a trained CHW and consists of three home-based visits with tailored print materials, text-messages delivered 2x/week, followed by monthly tailored print materials and phone calls during the last three months of the intervention. For in-home visits, the CHW will deliver a Motivational Interviewing session based on scripts developed in the R34. For phone calls, parents will receive a 30-minute Motivational Interviewing phone call to check in on goals and barriers and reinforce earlier concepts. For text messages, parents will be sent two times/week messages related to objectives targeted during that month's visit, such as parents setting good examples and giving children autonomy in eating. For print materials, parents will receive printed materials, highlighting nutrition and parental feeding guidance.
  Interventions: Behavioral: Home-Based Video and Motivational Interviewing Intervention
- Read Educate and Develop Youth (READY) Comparison (Active Comparator): As done in the R34, the comparison group will receive an attention contact control intervention about school readiness promotion adapted from R.E.A.D.Y. (Read Educate and Develop Youth) designed by the Michigan Department of Education (Refs). Families in the comparison arm will receive the same intervention components as the intervention arm, but these will be focused on child reading rather than nutrition. Parents will send a video of themselves reading with a child, receive 3 home visits and 48 text-messages as well as newsletters for each visit. Instead of receiving cooking materials during the second home visit, they will receive books to read with their children.
  Interventions: Behavioral: Read Educate and Develop Youth (READY) Comparison

INTERVENTIONS:
Behavioral: Home-Based Video and Motivational Interviewing Intervention — The intervention consists of three home-based visits, followed by phone calls during the last three months of the intervention. For each visit and phone call, participants will receive tailored print materials, and during the 6 months of the interventions, they will receive text messages 2x/week. The intervention will be delivered in English or Spanish by a bilingual Community Health Worker (CHW). The CHW will be hired to serve as MI counselors for the parents in the study, and will be in charge of delivering the MI in-home or telephone sessions. CHWs will be trained for 3 months, in Motivational Interviewing, study protocols, the use of video recordings, meal preparation, and cooking, and will undergo a MI certification process. During the sessions with the participants, the CHW will deliver semi-scripted MI sessions based on the scripts developed in the pilot study.
  Arms: Home-Based Video and Motivational Interviewing Intervention
Behavioral: Read Educate and Develop Youth (READY) Comparison — The comparison group will receive an attention contact control intervention about school readiness promotion adapted from R.E.A.D.Y. (Read Educate and Develop Youth) designed by the Michigan Department of Education. The intervention consists of three home-based visits, followed by phone calls during the last three months of the intervention. For each visit and phone call, participants will receive tailored print materials, and during the 6 months of the interventions, they will receive text messages 2x/week. The intervention will be delivered in English or Spanish by a bilingual Community Health Worker (CHW). Families will receive the same intervention components as the intervention, but about reading instead of nutrition.
  Arms: Read Educate and Develop Youth (READY) Comparison

SUMMARY:
The goal of this clinical trial is to test the ability of a home-based parental nutrition intervention to improve diet quality in preschool aged children within low-income, Latinx/Hispanic families. The main questions it aims to answer are:

* Does this enhanced intervention change children's diet quality?
* Does this enhanced intervention change parental feeding practices?
* Does this enhanced intervention change the availability of healthy foods in the home?

Participants will:

* Work with a support coach
* Have a home visit with a support coach once a month, for three months
* Have a phone call with a support coach once a month, for three months
* Receive written materials and text messages over the six months

Researchers will compare a control group receiving different written materials and messages to see if the enhanced intervention changes diet quality in children.

DETAILED DESCRIPTION:
Investigators will build on the recently completed R34 (R34HL140229) that developed and pilot-tested the feasibility, acceptability, and preliminary efficacy of a novel home-based intervention to improve the diet quality and home food environment of low-income, ethnically diverse preschool children (87% Latinx). Despite the study occurring during COVID-19, the intervention delivery was feasible and acceptable to participants and achieved encouraging improvements in children's diet quality and positive food parenting practices. For the proposed research the investigators will build upon lessons learned in the pilot to evaluate the efficacy of the novel Strong Families intervention to improve food parenting practices, home food environment, parent, and children's diet quality in a fully powered randomized controlled trial (RCT) with 257 families of a 2-5-year-old child. The intervention will include:

* Home visits by a community health worker (CHW) trained in brief motivational interviewing; screening for social-determinants of health and connecting families to federal/state/local resources; in-home cooking demonstrations to prepare a meal involving their child; feedback about a family meal-time video
* Text-messages
* Tailored materials/messages
* CHW phone calls

These strategies are expected to connect families to community systems, increase parental knowledge, self-efficacy, and motivation for serving easy, inexpensive healthy foods leading to increased child exposure to more healthy and varied foods, improvements in parental feeding practices and ultimately, improvements in child diet quality. The RCT will include baseline, 6 & 12-month measurements to test the following aims:

* Aim 1: Improve the dietary intakes of 2-5-year-old children
* Aim 2: Improve food parenting practices
* Aim 3. Improve the availability of healthy foods in the home

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Self-identity as Latinx/Hispanic
* Speak English or Spanish
* Be the primary caregiver of a child between 2- 5 years of age
* Live with the child most of the time
* Eat a minimum of three evening meals per week with the child
* Not have participated in the R34 study
* Have a smart phone
* Be willing to have a meal video recorded in the home

Exclusion Criteria:

* A doctor or WIC provider has told them that their child was underweight in the past 6 months
* The child has a diagnosed feeding disorder or dietary restriction that impacts how they eat

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 257 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Child Diet Quality | 2-24-Hour Recalls at Baseline and 2-24-Hour Recalls at 6-Month follow-up
  Caloric and macronutrient intake will be averaged over two dietary recalls. Caloric and macronutrient intake will be averaged over the two recalls. Healthy Eating Index (HEI)-2015 components (total fruit, whole fruit, total vegetable, dark green and orange vegetables and legumes, total grain, whole grain, milk, meat and beans, saturated fat, sodium, added sugars, and solid fats) are assessed per 1000 kcal to provide a density-based score except for saturated fats and added sugars with are % of energy. Component scores are then summed to provide a total HEI score.
Child's Dermal Carotenoids | Baseline, 6-Month Follow-up
  The Veggie Meter device will provide an objective, non-invasive and quick measure reflecting fruit and vegetable intake. This device uses reflection spectroscopy to detect the level of carotenoids in human skin. Three measures (10 seconds each spaced by 30-seconds) will be taken and averaged. Scores range from 0 to 800 with higher scores indicating greater fruit and vegetable intake.

SECONDARY OUTCOMES:
Food Parenting Practices | Baseline, 6-Month Follow-up
  Food parenting practices will be measured by the Food Parenting Inventory. Investigators will measure pre-post changes to 8 subscales: 1) child involvement in food preparation; 2) responsiveness to child's fullness cues; 3) encourage exploration of new foods; 4) repeated presentation of new foods; 5) regular timing of meals and snacks; 6) encourage try new foods; 7) inconsistent mealtimes; 8) food as a reward; and the Healthy Eating Guidance subscale of the Comprehensive Feeding Practices Questionnaire. All of the items are rated on a 5-point Likert scale ranging from never-always and disagree-agree. Higher subscale scores indicate greater use of that practice.
Availability of Healthy Foods in the Home | Baseline, 6-Month Follow-up
  The Home Food Inventory (HFI) will be used to assess a range of available foods in the home environment. Research staff will inventory the foods in the kitchen. The HFI includes 13 food categories (e.g., cheese, milk/dairy, F&V), whether F&V were fresh, canned/jarred, frozen, or dried, and two categories on food accessibility. HFI items are listed in a checklist format with yes/no options.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Tovar, PhD MPH, Principal Investigator — Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tovar A, Bouchard KL, Moore AM, Perry M, Lurssen I, Arriola Carnicelli L, Sanchez Contreras A, Risica P, von Ash T, Savage JS, Dunsiger S, Gans K. Strong Families Start at Home/Familias Fuertes Comienzan en Casa-Improving Child Diet Quality and Parental Feeding Practices: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Sep 10;14:e73923. doi: 10.2196/73923. PMID 40929716

DOCUMENTS (1):
  • Informed Consent Form (2022-09-07): https://cdn.clinicaltrials.gov/large-docs/88/NCT06099288/ICF_000.pdf